CLINICAL TRIAL: NCT00611169
Title: The Effects of Facilitated Percutaeous Coronary Intervention Compared to Primary Percutaneous Coronary Intervention in Patients With ST-Segment Elevation Acute Myocardial Infarction
Brief Title: The Effects of Facilitated Percutaeous Coronary Intervention in Acute Myocardial Infarction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: HC Gwon, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2005-09-007-001
Record Dates: First submitted 2008-01-27; First posted 2008-02-08 (Estimated); Last update posted 2008-02-08 (Estimated); Status verified 2007-08

CONDITIONS: Acute Myocardial Infarction
Keywords: Angioplasty, Transluminal, Percutaneous Coronary; tirofiban; Magnetic Resonance Imaging; Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction | interventions — Tirofiban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Aspirin, clopidogrel, unfractionated heparin plus tirofiban infusion at high bolus dose
  Interventions: Drug: tirofiban
- 2 (No Intervention): Aspirin, clopidogrel, unfractionated heparin

INTERVENTIONS:
Drug: tirofiban — tirofiban (25 μg/kg bolus and 0.15 μg/kg/min maintenance infusion for 24 hours)
  Arms: 1

SUMMARY:
The purpose of this study to investigate whether the administration of high-dose tirofiban before primary PCI could reduce myocardial infarct size, using analysis of contrast-enhanced magnetic resonance imaging.

ELIGIBILITY:
Inclusion Criteria:

* presence of chest pain for more than 30 minutes but less than 12 hours after symptom onset
* ST-segment elevation more than 1 mm in two or more contiguous leads or presumably a new-onset left bundle branch blockage

Exclusion Criteria:

* hemodynamic instability
* history of MI
* old age > 80years
* Patients with bleeding diathesis (coagulopathy, thrombocytopenia or platelet dysfunction, Gastrointestinal or genitourinary bleeding within the prior 3 months)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-01; Primary Completion 2007-02 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Infarct size and its transmural extent using MRI | within the first 30 days after index procedure

SECONDARY OUTCOMES:
pre-PCI thrombolysis in myocardial infarction grade, post-PCI myocardial blush grade, ST-segment resolution on electrocardiography, and left ventricular ejection fraction on echocardiography | at 6 month after index procedure

CONTACTS AND LOCATIONS:
Overall Officials: Hyeon-Cheol Gwon, MD, PhD, Principal Investigator — Samsung Medical Center